CLINICAL TRIAL: NCT05947006
Title: Study of the Impact of the Setting up of a Pediatric Nurse's Consultation on Parental Anxiety During a Febrile Convulsion in Children
Brief Title: Study of the Impact of a Pediatric Nurse's Consultation on Parental Anxiety During a Febrile Convulsion in Children
Acronym: CONSULFE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigator changed departments, parents refused to participate in the study
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC31/22/0484
Record Dates: First submitted 2023-06-19; First posted 2023-07-14 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Febrile Seizure
Keywords: anxiety; fever; convulsion; seizure; children
MeSH Terms: conditions — Seizures, Febrile; Anxiety Disorders; Fever; Seizures | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Prospective, controlled, non-randomized single-center pilot study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard care (Active Comparator): Patients in this arm will receive the standard care stablished in the emergency room after a febrile seizure
  Interventions: Other: Standard care
- CONSULFE Consultation (Experimental): Patients in this arm will receive a consultation managed by the pediatric nurse (CONSULFE)
  Interventions: Other: CONSULFE consultation

INTERVENTIONS:
Other: Standard care — Patients in this arm will receive the standard care stablished in the emergency room after a febrile seizure, consisting of a medical assessment of the child, followed by 6 hours of supervision of the child and his parent in the waiting room, a reassessment of the child by the doctor, and finally they can return home
  Arms: Standard care
Other: CONSULFE consultation — In addition to the standard care, patients in this arm will receive a consultation managed by the pediatric nurse (CONSULFE) during the 6 hour supervision time in the waiting room
  Other Names: Consultation managed by the pediatric nurse
  Arms: CONSULFE Consultation

SUMMARY:
Febrile seizures are considered a very common syndrome presented in the pediatric emergency room. Witnessing these seizures may can cause anxiety in parents and generate them psychological sequelae such as major depressive disorder in the short term, or sleep disorders in the long term.

An appropriate care for parents must be put in place in the emergency department, with the objective of improving their knowledge of this pathology and its care, and thus to reduce their anxiety and prevent potential inappropriate or even deleterious behavior and maneuvers towards the child.

DETAILED DESCRIPTION:
Febrile seizures occupy a large place in pediatric practice in the emergency room, their prevalence varies between 3 and 8% in children under 7 years old, hence the notion of a very common syndrome.

When parents witness this event, they can experience it as terrifying, and which can alone cause anxiety and generate psychological sequelae. In the literature, it is described that a third of the parents present a major depressive disorder after the event and a third of the parents still describe sleep disorders after one year.

After the arrival at the pediatric emergency room following the febrile seizure, the priority is given to the care of the child and parents are given succinct medical information. Due to parental anxiety, which may still be significant at this time, this information may not be understood. All of this can make the parent's level of knowledge about this pathology and its management low, potentially leading to future behaviors and maneuvers (such as shaking) that are inappropriate or even harmful to the child.

A different course with appropriate care for parents must be put in place in the emergency department, with the objective of improving their knowledge of this pathology, its care and to reduce parent's anxiety. This is why the CONSULFE childcare consultation is proposed in this research.

ELIGIBILITY:
Inclusion Criteria:

* Participant being an adult parent who attended the febrile seizure of their child aged 1 to 5, episode lasting less than 15 minutes occurring within 24 hours
* Participant having signed the free and informed consent
* Affiliation to a social security scheme

Exclusion Criteria:

* Parent who already has experience of febrile seizures in one of the siblings
* Parent of a child with a convulsive or neurological history
* Non-French speaking parents
* Parent with a diagnosed psychiatric illness
* Parent benefiting from a legal protection measure
* Parent participating in a study related to the management of anxiety

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2024-04-22 (Actual); Primary Completion 2025-03-04 (Actual); Study Completion 2025-03-04 (Actual)

PRIMARY OUTCOMES:
Level of anxiety | Baseline and 6 hours after the intervention
  Change in the level of anxiety felt at the beginning and at the end of the visit to the emergency room by parents during standard treatment vs parents following the CONSULFE consultation. The level of anxiety is measured with the State-Trait Anxiety Inventory (STAI), with a minimum value of 20, meaning no or low anxiety, and a maximum value of 80, meaning high anxiety.

SECONDARY OUTCOMES:
Parent's level of anxiety upon arrival on the emergency room | Baseline
  Level of anxiety measured by the State-Trait Anxiety Inventory (STAI), with a minimum value of 20, meaning no or low anxiety, and a maximum value of 80, meaning high anxiety.
Parent's socio-economic position | Baseline
  Socio-economic position of parents measured by their level of study
Parent's level of anxiety at the departure of the emergency room | 6 hours after the intervention
  Level of anxiety measured by the State-Trait Anxiety Inventory (STAI), with a minimum value of 20, meaning no or low anxiety, and a maximum value of 80, meaning high anxiety.
Satisfaction of parents with intervention | 6 hours after the intervention
  Satisfaction with the intervention will be measured using a satisfaction questionnaire with values between 1 and 4, 1 meaning completely satisfied, and 4 meaning not satisfied
Long term parent's level of anxiety | 1 month after the intervention
  Level of anxiety measured by the State-Trait Anxiety Inventory (STAI), with a minimum value of 20, meaning no or low anxiety, and a maximum value of 80, meaning high anxiety.
Long term parent's level of post-traumatic stress | 1 month after the intervention
  Post-traumatic stress (PTSD) measured by the IMPACT OF EVENTS SCALE-Revised (IES-R), with a minimum value of 0, meaning no PTSD, and a maximum value of 88, meaning PTSD is high enough to suppress your immune system's functioning
Cost of the intervention | 1 month after the intervention
  The costs will be estimated according to two perspectives : from the hospital point of view (time spent by the childcare nurse), and from the health insurance point of view (number of consultations and visits to the emergency room)

CONTACTS AND LOCATIONS:
Overall Officials: Alex BRIGAND, Principal Investigator — University Hospital, Toulouse
Locations (1):
- CHU Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tison-Chambellan C, Fine A, Cances C, Chaix Y, Claudet I. [Anthropological approach to current parental perceptions of children's seizures]. Arch Pediatr. 2013 Oct;20(10):1075-82. doi: 10.1016/j.arcped.2013.07.001. Epub 2013 Aug 7. French. PMID 23932660
- [Background] Balslev T. Parental reactions to a child's first febrile convulsion. A follow-up investigation. Acta Paediatr Scand. 1991 Apr;80(4):466-9. doi: 10.1111/j.1651-2227.1991.tb11883.x. PMID 2058397
- [Background] Kolahi AA, Tahmooreszadeh S. First febrile convulsions: inquiry about the knowledge, attitudes and concerns of the patients' mothers. Eur J Pediatr. 2009 Feb;168(2):167-71. doi: 10.1007/s00431-008-0724-z. Epub 2008 May 7. PMID 18461360
- [Background] Paul SP, Rogers E, Wilkinson R, Paul B. Management of febrile convulsion in children. Emerg Nurse. 2015 May;23(2):18-25. doi: 10.7748/en.23.2.18.e1431. PMID 25952398
- [Background] Smith DK, Sadler KP, Benedum M. Febrile Seizures: Risks, Evaluation, and Prognosis. Am Fam Physician. 2019 Apr 1;99(7):445-450. PMID 30932454
- [Background] Walsh A, Edwards H, Fraser J. Influences on parents' fever management: beliefs, experiences and information sources. J Clin Nurs. 2007 Dec;16(12):2331-40. doi: 10.1111/j.1365-2702.2006.01890.x. Epub 2007 Apr 5. PMID 17419783
- [Background] Klotz KA, Ozcan J, Sag Y, Schonberger J, Kaier K, Jacobs J. Anxiety of families after first unprovoked or first febrile seizure - A prospective, randomized pilot study. Epilepsy Behav. 2021 Sep;122:108120. doi: 10.1016/j.yebeh.2021.108120. Epub 2021 Jun 15. PMID 34144460